CLINICAL TRIAL: NCT00179543
Title: Mechanisms and Therapeutic Effects of the Relaxation Response in Elderly Hypertensive Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2001-P-001727; CDC grant: H75-CCH-123424; CDC grant: H75-CCH-119124; CDC grant: R01 DP00039
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2006-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Behavioral: Relaxation response

SUMMARY:
The purpose of this study is to determine whether the relaxation response is more effective than attention control in reducing blood pressure and medication dosage in elderly adults with isolated systolic hypertension.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the relaxation response is more effective than health education training (attention control) in reducing systolic blood pressure and anti-hypertensive medication elimination in elderly adults with isolated systolic hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 55 years or older
* currently taking at least 2 anti-hypertensive medications
* systolic blood pressure between 140-159 mmHg
* diastolic blood pressure less than 90 mmHg
* read and understand English
* access to a telephone
* ability to attend all study visits

Exclusion Criteria:

* other cardiovascular disease
* major medical illness
* previous experience with any RR eliciting technique
* current use of:beta-agonist bronchodilators, systemic corticosteroids, anti-convulsants/psychotics, immunosuppressants, cytotoxic therapy, anabolic steroids, antidepressants (other than SSRIs), dicyclomine, bile acid binding resins, or sympathomimetic medication

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122
Dates: Start 2001-08

PRIMARY OUTCOMES:
Determine whether the relaxation response is more effective than a health education control in reducing blood pressure in elderly adults with isolated systolic hypertension.

SECONDARY OUTCOMES:
Evaluate whether the relaxation response is more effective than a health education control to safely reduce blood pressure medications in elderly adults with isolated systolic hypertension..

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Benson, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- BIDMC, Boston, Massachusetts, United States